CLINICAL TRIAL: NCT01688115
Title: Reduction of Preoperative Anxiety in Children: Clickamico Project 2nd Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Filippo Festini, Professor of Nursing, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IPAD2012
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Preoperative Anxiety
MeSH Terms: interventions — Videotape Recording; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procedure (Experimental)
  Interventions: Procedure: Video
- Standard Care (Active Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Video — The afternoon before the surgery session, a researcher will show to the child a video of the length of 6 minutes, using an I-pad. The video shows two clown doctors working constantly at Meyer Children's Hospital, which, through skits and gags, will tell the child how is an operating room and some devices and procedures used during the induction of anesthesia.
  Arms: Procedure
Other: Standard care — In this arm orally information will be given by the nurse of the ward only to the parents of the child. Any additional information or explanation will be given to the child
  Arms: Standard Care

SUMMARY:
The purpose of this study is to evaluate the efficacy of a video shown using an iPad, compared to a standard treatment, to reduce preoperative anxiety in children who have to undergo to elective surgery procedure

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 11
* No cerebral impairment or cognitive impairment
* Child and his/her family native speaker of Italian
* admission to the hospital at list one day before the sugery procedure
* presence of written consent of the parents to the study

Exclusion Criteria:

* age lower than 6 or upper than 11
* presence of cerebral impairment or cognitive impairment
* Child and his/her family are not native speaker of Italian
* absence of written consent of the parents to the study

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | perhaps 24 hours from child admission to surgery procedure
  Preoperative anxiety is measured using the "Modified Yale Preoperative Anxiety Scale (m-YPAS)"

REFERENCES:
- [Derived] Liguori S, Stacchini M, Ciofi D, Olivini N, Bisogni S, Festini F. Effectiveness of an App for Reducing Preoperative Anxiety in Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):e160533. doi: 10.1001/jamapediatrics.2016.0533. Epub 2016 Aug 1. PMID 27294708